CLINICAL TRIAL: NCT04362384
Title: Topical Endorectal Vietamin E Ovules for the Treatment of Grade 2 and 3 Hemorrhoids
Brief Title: Topical Vitamin E Ovules for the Treatment of Hemorrhoids
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Department of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Garcilaso 2020/2
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Bleeding Anal; Pain; Stings
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Pain; Bites and Stings | interventions — neomycin, prednisolone, surfen, trypsin-chymotrypsin drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Symptoms will be assessed by a nurse blinded to the prescribed treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin E ovules (Experimental): Endoanal Vitamin E ovules will be prescriped during 14 days
  Interventions: Drug: Vitamin E ovules
- Prednisolone ointment (Active Comparator): Endoanal Prednisolone ointment will be prescriped during 14 days
  Interventions: Drug: Prednisolone ointment

INTERVENTIONS:
Drug: Vitamin E ovules — Endoanal vitamin E ovules will be prescribed
  Arms: Vitamin E ovules
Drug: Prednisolone ointment — Endoanal Prednisolone ointment will be prescribed
  Arms: Prednisolone ointment

SUMMARY:
Patients with hemorrohoids grade II and III were included. Patients were randomized into 2 groups:

* Experimental group: Patients will receive a treatment with vitamin E ovules, which must be placed inside the annus
* Control group: Patients will receive a treatment with corticoid ointment, with endoanal application

Bleeding, pain and stinging will be evaluated 14 days after beginning the treatment.

DETAILED DESCRIPTION:
Patients with hemorrohoids grade II and III were included.

Patients were randomized into 2 groups:

* Experimental group: Patients will receive a treatment with vitamin E ovules, which must be placed inside the annus. 1 ovule must be inserted daily during 14 days.
* Control group: Patients will receive a treatment with prednisolone ointment, with endoanal application 3 times per day during 14 days.

Bleeding, pain and stinging will be evaluated 14 days after beginning the treatment. Quantification of pain will be performed following a visual analogic scale ranging from 0 (absence of symptoms) to 100 (unbearable symptoms).

ELIGIBILITY:
Inclusion Criteria:

* Grade II and III hemorrhoids

Exclusion Criteria:

* Grade I or IV hemorrhoids
* Patients with previous anal surgeries
* Patients having received previous pharmacological treatments for hemorrhoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
% of patients with Bleeding | 14 days after beginning the treatment
  The patient refers rectal bleeding during defecation (patients´self-report) or active bleeding is observed at rectal examination. The variable will be measured as present (1) or absent(0)

SECONDARY OUTCOMES:
Anal pain assessed by Visual Analogic Scale | 14 days after beginning the treatment
  The patients will be asked to quantify their perception of pain on a VAS, ranging from 0mm(absence of pain) to 100mm (unbearable pain)
% of patients with Stinging | 14 days after beginning the treatment
  The patient refers stinging sensation (patients´self-report) . The variable will be measured as present (1) or absent(0)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz Tovar Polo, Principal Investigator — Garcilaso Clinic